CLINICAL TRIAL: NCT02706145
Title: Changing the Narrative: Using Media to Shift Social Norms of Violence Among Youth in West Louisville
Brief Title: Using Media to Shift Social Norms of Violence Among Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Vanderbilt University (Other)
Responsible Party: Principal Investigator, Monica L. Wendel, Associate Professor, University of Louisville
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15.0910; 1U01CE002711 (NIH)
Record Dates: First submitted 2016-02-23; First posted 2016-03-11 (Estimated); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Violence
Keywords: social norms; youth violence; media

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (West Louisville) (Experimental): This group will be exposed to the social norming campaign via traditional, mass, and social media over the three-year intervention period.
  Interventions: Other: Social norming campaign
- Control Group (East Nashville) (No Intervention): This group will serve as the control group, and measures of social norms and attitudes toward violence will be compared between this group and the intervention group.

INTERVENTIONS:
Other: Social norming campaign — community-level, three-year social norming campaign, using traditional and emerging media, aimed at changing norms of violence among youth 10-24
  Arms: Intervention Group (West Louisville)

SUMMARY:
The project will utilize a quasi-experimental design to examine the effectiveness of a community-level, three-year social norming campaign aimed at changing norms of violence among youth 10-24, with West Louisville (WL) as the intervention community and East Nashville, Tennessee as the control community. The project will address the following research questions (RQs):

RQ1: To what extent is a social norming campaign effective in changing the descriptive and injunctive norms of violence among youth in WL?

RQ2: To what extent are the descriptive and injunctive norms of violence among youth in WL related to violent behavior (by type)?

RQ3: To what extent is a social norming campaign effective in reducing population rates of youth violence in WL?

RQ4: Which forms of media are most effective in reaching youth of different ages with campaign messages?

RQ5: How is community readiness related to implementation of a community-level social norming campaign?

RQ6: How is community capacity related to implementation of a community-level social norming campaign?

RQ7: How does community capacity to address youth violence change over time with the implementation of a community-level social norming campaign?

RQ8: To what extent is a social norming campaign cost-effective in reducing incidents of serious violence among youth?

DETAILED DESCRIPTION:
The Center of Excellence in Youth Violence Prevention at the University of Louisville (UofL) School of Public Health & Information Sciences capitalizes on a specific window of opportunity-where there is currently alignment of a public consciousness of the issue of youth violence, the availability of expertise to implement a feasible intervention, and substantial political will across community sectors to address the issue. This provides an ideal context for the creation of the UofL Center for Youth Violence Prevention, allowing us to partner with residents and organizations in West Louisville (WL) to develop, implement, and evaluate a community-level intervention to reduce youth violence. To this end, we plan to achieve five specific aims:

AIM 1: Strengthen the infrastructure to support youth violence prevention research and practice at the University of Louisville.

AIM 2: Develop, implement and evaluate a community-level social norming campaign to change the norms of violence among youth in West Louisville using mass and social media.

AIM 3: Document the development and implementation of the social norming campaign to improve replication and scalability in other settings or communities.

AIM 4: Evaluate the relationship between community readiness, community capacity, and the implementation of the community-level social norming campaign.

AIM 5: Facilitate knowledge translation and dissemination initiatives to relevant audiences (i.e., community, local organizations and leaders, youth violence prevention researchers and practitioners, academic peers, and policy-makers) that produce actionable community- and policy-level approaches.

ELIGIBILITY:
Inclusion Criteria:

* youth between 10 and 24 years of age who reside in one of the nine neighborhoods of West Louisville or in the comparison site of East Nashville

Exclusion Criteria:

* individuals outside the age range (i.e., younger than 10 or older than 24) or who do not live in the intervention or comparison communities

Ages: 10 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 8037 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of youth who report descriptive norms that promote violence as measured by our school survey | up to 60 months
  Survey will assess population level changes in descriptive norms among youth in the intervention group related to violence compared to control group
Proportion of youth who report injunctive norms that promote violence as measured by our school survey | up to 60 months
  Survey will assess population level changes in injunctive norms among youth in the intervention group related to violence compared to youth in the control group
Proportion of youth who engaged in violent behavior in the past 12 months as measured by our school survey | up to 60 months
  Youth engagement in violent behavior (by type of violence)
Community rates of violence involving youth 10-24 aggregated by police department, emergency department, and school district records | up to 60 months
  Community-level rates of youth violence (by type of violence)

CONTACTS AND LOCATIONS:
Overall Officials: Monica L Wendel, DrPH, Principal Investigator — University of Louisville School of Public Health; Maury Nation, PhD, Principal Investigator — Vanderbilt University
Locations (2):
- United States (2):
  - University of Louisville School of Public Health & Information Sciences, Louisville, Kentucky
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Will share data, but nothing with identifiers

REFERENCES:
- [Background] Castle B, Wendel M, Kerr J, Brooms D, Rollins A. Public Health's Approach to Systemic Racism: a Systematic Literature Review. J Racial Ethn Health Disparities. 2019 Feb;6(1):27-36. doi: 10.1007/s40615-018-0494-x. Epub 2018 May 4. PMID 29729001
- [Background] Wendel ML, Jones G Jr. Equity for Whom? The Example of Qualified Opportunity Zones. Am J Public Health. 2020 Mar;110(3):280-281. doi: 10.2105/AJPH.2019.305532. No abstract available. PMID 32023101
- [Background] Wendel ML. Commentary: Racism is a Public Health Emergency. Fam Community Health. 2020 Oct/Dec;43(4):255-256. doi: 10.1097/FCH.0000000000000281. No abstract available. PMID 32826736
- [Result] Castle B, Wendel M, Kelly Pryor BN, Ingram M. Assessing Community Leadership: Understanding Community Capacity for Health Improvement. J Public Health Manag Pract. 2017 Jul/Aug;23 Suppl 4 Suppl, Community Health Status Assessment:S47-S52. doi: 10.1097/PHH.0000000000000587. PMID 28542064
- [Result] Golden TL, Wendel ML. Public Health's Next Step in Advancing Equity: Re-evaluating Epistemological Assumptions to Move Social Determinants From Theory to Practice. Front Public Health. 2020 May 7;8:131. doi: 10.3389/fpubh.2020.00131. eCollection 2020. PMID 32457863
- See also: Campaign Website — http://pridepeaceprevention.org